CLINICAL TRIAL: NCT02995915
Title: Mobile Contingency Management for Concurrent Abstinence From Alcohol and Smoking
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00062101
Record Dates: First submitted 2016-12-14; First posted 2016-12-19 (Estimated); Results first posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Smoking Cessation; Alcohol Drinking
MeSH Terms: conditions — Smoking Cessation; Alcohol Drinking | interventions — Nicotine Replacement Therapy; Nicotine Chewing Gum; Transdermal Patch; Nebulizers and Vaporizers; Bupropion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tele-health Mobile Contingency Management Intervention (Experimental): This arm includes a proactive tele-health intervention that combines evidence-based telephone cognitive behavioral treatment for alcohol and smoking cessation, a tele-medicine clinic for access to smoking cessation pharmacotherapy (including nicotine replacement therapy and bupropion), and mobile contingency management treatment administered via a smart-phone based application (mobile CM).
  Interventions: Other: Nicotine Replacement Therapy; Drug: Bupropion; Behavioral: Cognitive Behavioral Treatment; Behavioral: Mobile Contingency Management
- Tele-health for Alcohol and Smoking Cessation (Active Comparator): This arm includes a proactive tele-health intervention that will provide controls for therapist, medication, time and attention effects. The tele-health intervention provides the same evidence-based telephone CBT for alcohol and smoking cessation, and tele-medicine clinic for access to smoking cessation pharmacotherapy as in the mCM intervention, but does not include mCM. Instead, participants will receive monetary compensation for each assessment, regardless of abstinence.
  Interventions: Other: Nicotine Replacement Therapy; Drug: Bupropion; Behavioral: Cognitive Behavioral Treatment; Behavioral: Mobile Monitoring

INTERVENTIONS:
Other: Nicotine Replacement Therapy — Participants will be prescribed NRT patch and one nicotine rescue method (e.g., nicotine gum, lozenge, inhaler) for use during the post-quit phase of the study. Participants will be given the choice between nicotine gum or nicotine lozenge, and will be instructed to use the rescue method as needed to reduce cigarette cravings
  Other Names: nicotine gum, patch, inhaler, and/or lozenge
Drug: Bupropion — All participants who are medically eligible will be prescribed bupropion, which they will start two weeks prior to their quit day. Dosage will be 150 mg/daily for days 1-7 and 300 mg/daily (administered in two daily doses) until the 6-month follow-up.
  Other Names: Zyban
Behavioral: Cognitive Behavioral Treatment — Participants will receive 4 60-minute sessions of CBT telephone counseling for alcohol and smoking cessation.
  Other Names: CBT
Behavioral: Mobile Contingency Management — Participants will be asked to provide video recordings of themselves taking carbon monoxide readings in order to confirm smoking abstinence, and breathalyzer to confirm abstinence from alcohol. Participants are asked to upload these videos to the study's secured server, and are provided monetary reward for videos that suggest smoking abstinence and alcohol abstinence.
  Other Names: mobile CM, mCM
  Arms: Tele-health Mobile Contingency Management Intervention
Behavioral: Mobile Monitoring — Participants will be asked to provide video recordings of themselves taking carbon monoxide readings and breathalyzer. Participants are asked to upload these videos to the study's secured server, and are provided monetary reward for providing the video recordings, regardless of abstinence.
  Arms: Tele-health for Alcohol and Smoking Cessation

SUMMARY:
Alcohol misuse and smoking constitute two of the three leading preventable causes of death in the United States. The purpose of this research study is to develop an intervention designed to help people stop drinking alcohol and stop smoking at the same time.

DETAILED DESCRIPTION:
Alcohol misuse and smoking constitute two of the three leading preventable causes of death in the United States. Reluctance to treat tobacco dependence among those with AUD is misguided as recent research suggests smoking cessation treatment can be effective, does not increase risk of relapse to alcohol, and may even improve rates of sobriety. There is strong evidence for the short-term efficacy for alcohol misuse and smoking of contingency management (CM). It is an intensive behavioral therapy that provides incentives (vouchers, money) to individuals misusing substances contingent upon objective evidence from drug use. Implementation of CM has been limited because of the need to verify abstinence multiple times daily using clinic based monitoring. The investigators recently developed a smart-phone application which allows a patient to video themselves several times daily while using a small CO monitor and to transmit the data to a secure server which has made the use of CM for outpatient smoking cessation portable and feasible. This mobile CM (mCM) approach paired with cognitive-behavioral counseling and pharmacological smoking cessation aids has been effective in reducing smoking.

Thus, the purpose of this project is to develop a combined alcohol and smoking mCM intervention. The intervention will be developed in two successive cohorts of five participants, who will provide information on treatment acceptability and feasibility. A third cohort of participants (n=45) will participate in a randomized clinical trials to further examine feasibility and efficacy. The long term goal is to develop mCM procedures that will be used as part of a multi-component intervention to concurrently and effectively treat both alcohol misuse and smoking. As part of this project, the investigators will develop a multi-component telehealth alcohol and smoking mCM intervention. It will include mCM, cognitive-behavioral phone counseling, and standard smoking cessation pharmacotherapy. The work proposed in these aims will provide the first step toward implementation of an innovative approach that builds upon the power of mHealth technology to reduce the prevalence of both alcohol misuse and smoking.

ELIGIBILITY:
Inclusion Criteria:

* currently meet criteria for DSM-5 mild to moderate alcohol use disorder (meeting 2-5 criteria for AUD)
* have been engaging in hazardous drinking over the past month, defined as either exceeding a mean of 14 standard drinks/wk for men, 7 drinks/wk for women; or by consuming >5 on at least one occasion in the last month for men, >4 drinks on at least one occasion in the last month for women
* currently smoke >10 cigarettes a day, and have smoked for at least one year
* can speak and write fluent conversational English
* are willing to make an attempt to quit both alcohol and smoking

Exclusion Criteria:

* are expected to have unstable medication regimen during the study
* are currently receiving non-study behavioral treatment for alcohol use disorder or smoking
* have severe alcohol use disorder (meeting >6 criteria for AUD or having alcohol withdrawal symptom criterion)
* have AUD that is in early remission, with no symptoms evident over the past month
* have experienced myocardial infarction in past 6 months
* contraindication to nicotine replacement therapy with no medical clearance to participate in the study
* use other forms of nicotine such as cigars, pipes, or chewing tobacco
* are currently pregnant
* have a primary psychotic disorder or current manic episode
* have had substance use disorder (other than alcohol or nicotine) in the preceding 3 months
* are currently imprisoned or in psychiatric hospitalization

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-11; Primary Completion 2020-03-02 (Actual); Study Completion 2020-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric A. Dedert, Ph.D., Principal Investigator — Study Principal Investigator
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Tele-health Mobile Contingency Management Intervention: This arm includes a tele-health intervention that combines evidence-based telephone cognitive behavioral treatment for alcohol and smoking cessation, smoking cessation pharmacotherapy (including nicotine replacement therapy and bupropion), and mobile contingency management treatment administered via a smart-phone based application (mobile CM).
  Nicotine Replacement Therapy: Participants will be prescribed NRT patch and one nicotine rescue method (e.g., nicotine gum, lozenge, inhaler) for use during the post-quit phase of the study. Participants will be given the choice between nicotine gum or lozenge, and will be instructed to use the rescue method as needed to reduce cigarette cravings
  Bupropion: All medically eligible participants will be prescribed bupropion, which they will start two weeks prior to their quit day. Dosage will be 150 mg/daily for days 1-7 and 300 mg/daily (administered in two daily doses) until the 6-month follow-up.
  Cognitive Behavioral Treatment: Participants will receive 4 60-minute sessions of CBT telephone counseling for alcohol and smoking cessation.
  Mobile Contingency Management: Participants will be asked to provide video recordings of themselves taking carbon monoxide readings in order to confirm smoking abstinence, and breathalyzer to confirm abstinence from alcohol. Participants are provided monetary reward for videos that suggest smoking abstinence and alcohol abstinence.
- Tele-health for Alcohol and Smoking Cessation: This arm includes a tele-health intervention that will provide controls for therapist, medication, time and attention effects. The tele-health intervention provides the same evidence-based telephone CBT for alcohol and smoking cessation, and smoking cessation pharmacotherapy as in the mCM intervention, but does not include mCM. Instead, participants receive monetary compensation for each assessment, regardless of abstinence.
  Nicotine Replacement Therapy: Participants will be prescribed NRT patch and one nicotine rescue method (e.g., nicotine gum, lozenge, inhaler) for use during the post-quit phase of the study. Participants will be given the choice between nicotine gum or lozenge, and will be instructed to use the rescue method as needed to reduce cigarette cravings
  Bupropion: medically eligible participants will be prescribed bupropion, which they will start two weeks prior to their quit day. Dosage will be 150 mg/daily for days 1-7 and 300 mg/daily (administered in two daily doses) until the 6-month follow-up.
  Cognitive Behavioral Treatment: Participants will receive 4 60-minute sessions of CBT telephone counseling for alcohol and smoking cessation.
  Mobile Monitoring: Participants will be asked to provide video recordings of themselves taking carbon monoxide readings and breathalyzer. Participants are asked to upload these videos to the study's secured server, and are provided monetary reward for providing the video recordings, regardless of abstinence.
Period: Overall Study
Arm/Group | Tele-health Mobile Contingency Management Intervention | Tele-health for Alcohol and Smoking Cessation
Started | 30 | 15
Completed | 30 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tele-health Mobile Contingency Management Intervention | Tele-health for Alcohol and Smoking Cessation | Total
Number analyzed (Participants) | 30 | 15 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.77 (11.39) | 42.67 (11.46) | 42.73 (11.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 24 | 12 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 30 | 15 | 45
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 11 | 32
  White | 7 | 2 | 9
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 15 | 45

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Self-report Prolonged Abstinence From Smoking
Description: Participants will be asked to report on smoking since two weeks past quit date
Time Frame: 6 month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Tele-health Mobile Contingency Management Intervention | Tele-health for Alcohol and Smoking Cessation
Number analyzed (Participants) | 30 | 15
Participants | 3 | 0

2. Primary Outcome: Number of Participants Whose Prolonged Abstinence From Smoking is Bio-verified
Description: Self-reported prolonged abstinence (primary outcome) will be verified by cotinine assay. Saliva samples will be collected from participants who self-report prolonged abstinence.
Time Frame: 6 month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Tele-health Mobile Contingency Management Intervention | Tele-health for Alcohol and Smoking Cessation
Number analyzed (Participants) | 30 | 15
Participants | 2 | 0

3. Primary Outcome: Number of Participants Who Self-report Prolonged Abstinence From Alcohol Use
Description: Participants will be asked to report on alcohol use since two weeks past quit date
Time Frame: 6 month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Tele-health Mobile Contingency Management Intervention | Tele-health for Alcohol and Smoking Cessation
Number analyzed (Participants) | 30 | 15
Participants | 4 | 0

4. Primary Outcome: Number of Participants Whose Prolonged Abstinence From Alcohol is Bio-verified
Description: Self-reported prolonged abstinence will be verified by breathalyzer. Breathalyzer data will be collected from participants who self-report prolonged abstinence.
Time Frame: 6 month follow-up
Population: This subset of participants self-reported prolonged abstinence from alcohol.
Measure: Count of Participants; unit: Participants
Arm/Group | Tele-health Mobile Contingency Management Intervention | Tele-health for Alcohol and Smoking Cessation
Number analyzed (Participants) | 4 | 0
Participants | 4 | 0

5. Primary Outcome: Number of Participants Who Self-report Prolonged Dual Abstinence From Both Smoking and Alcohol
Description: Participants will be asked to report on smoking and alcohol use since two weeks past quit date
Time Frame: 6 month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Tele-health Mobile Contingency Management Intervention | Tele-health for Alcohol and Smoking Cessation
Number analyzed (Participants) | 30 | 15
Participants | 1 | 0

6. Primary Outcome: Number of Participants Whose Prolonged Dual Abstinence From Alcohol and Smoking is Bio-verified
Description: Self-reported prolonged abstinence from smoking will be verified by cotinine assay. Saliva samples will be collected from participants who self-report prolonged abstinence.Self-reported prolonged abstinence will be verified by breathalyzer. Breathalyzer data will be collected from participants who self-report prolonged abstinence.
Time Frame: 6 month follow-up
Population: This subset of participants self-reported dual abstinence from alcohol use and smoking.
Measure: Count of Participants; unit: Participants
Arm/Group | Tele-health Mobile Contingency Management Intervention | Tele-health for Alcohol and Smoking Cessation
Number analyzed (Participants) | 1 | 0
Participants | 1 | 0

7. Secondary Outcome: Number of Participants Who Self-report 7 Day Point Prevalence Abstinence From Smoking
Description: 7-day point prevalence abstinence is defined as no smoking in the prior 7 days.
Time Frame: 6 month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Tele-health Mobile Contingency Management Intervention | Tele-health for Alcohol and Smoking Cessation
Number analyzed (Participants) | 30 | 15
Participants | 6 | 2

8. Secondary Outcome: Number of Participants Who Report 30 Day Point Prevalence Abstinence From Smoking
Description: 30-day point prevalence abstinence is defined as no smoking in the prior 30 days
Time Frame: 6 month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Tele-health Mobile Contingency Management Intervention | Tele-health for Alcohol and Smoking Cessation
Number analyzed (Participants) | 30 | 15
Participants | 5 | 1

9. Secondary Outcome: Change in the Proportion of Days in Which Consumed Alcohol Compared to Pre-quit Use
Description: Participants will self-report number of days drank alcohol in the past 30 days and this will be compared to self-reported number of days drank alcohol in 30 days prior to quit.
Time Frame: 6 month follow-up
Measure: Mean (Standard Deviation); unit: drinking days per month
Arm/Group | Tele-health Mobile Contingency Management Intervention | Tele-health for Alcohol and Smoking Cessation
Number analyzed (Participants) | 30 | 15
drinking days per month | -9.67 (9.68) | -10.3 (10.69)

10. Secondary Outcome: Change in the Number of Standard Alcoholic Beverages Consumed Per Week Compared to Pre-quit Use
Description: Participants will self-report number of alcoholic beverages consumed in past 7 days and this will be compared to self-reported number of alcoholic beverages consumed in 7 days prior to quit.
Time Frame: 6 month follow-up
Measure: Mean (Standard Deviation); unit: drinks per week
Arm/Group | Tele-health Mobile Contingency Management Intervention | Tele-health for Alcohol and Smoking Cessation
Number analyzed (Participants) | 30 | 15
drinks per week | -7.53 (17.54) | -13.9 (17.72)

11. Secondary Outcome: Change in the Number of Heavy Drinking Episodes Compared to Pre-quit Use
Description: Participants will self-report number of heavy drinking episodes in the past 30 days and this will be compared to self-reported number of heavy drinking episodes in 30 days prior to quit.
Time Frame: 6 month follow-up
Measure: Mean (Standard Deviation); unit: heavy drinking episodes
Arm/Group | Tele-health Mobile Contingency Management Intervention | Tele-health for Alcohol and Smoking Cessation
Number analyzed (Participants) | 30 | 15
heavy drinking episodes | -9.22 (10.22) | -11.00 (9.61)

12. Secondary Outcome: Number of Participants Who Are Able to Achieve Recommended Drinking Limits (i.e., Less Than or Equal to 14 Drinks Per Week and Fewer Than 5 Drinks Per Day for Men; Less Than or Equal to 7 Days Per Week and Less Than 4 Drinks Per Day for Women)
Description: Participants will be asked to report on alcohol use in past week
Time Frame: 6 month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Tele-health Mobile Contingency Management Intervention | Tele-health for Alcohol and Smoking Cessation
Number analyzed (Participants) | 30 | 15
Participants | 16 | 8

13. Secondary Outcome: Number of Participants Who Self-report Prolonged Abstinence From Alcohol Use
Description: Participants will be asked to report on alcohol use since two weeks past quit date
Time Frame: 6 week follow-up (i.e., end of treatment visit)
Measure: Count of Participants; unit: Participants
Arm/Group | Tele-health Mobile Contingency Management Intervention | Tele-health for Alcohol and Smoking Cessation
Number analyzed (Participants) | 30 | 15
Participants | 14 | 3

14. Secondary Outcome: Number of Participants Whose Prolonged Abstinence From Alcohol is Bio-verified
Description: as for outcome 4
Time Frame: 6 week follow-up (i.e., end of treatment visit)
Measure: Count of Participants; unit: Participants
Arm/Group | Tele-health Mobile Contingency Management Intervention | Tele-health for Alcohol and Smoking Cessation
Number analyzed (Participants) | 30 | 15
Participants | 13 | 1

15. Secondary Outcome: Change in Number of Average Cigarettes Smoked Per Day
Description: Participants will self-report average number of cigarettes smoked in the past week and this will be compared to self-reported number of smoked in the week prior to quit.
Time Frame: 6 month follow-up
Measure: Mean (Standard Deviation); unit: cigarettes per day
Arm/Group | Tele-health Mobile Contingency Management Intervention | Tele-health for Alcohol and Smoking Cessation
Number analyzed (Participants) | 30 | 15
cigarettes per day | -8.56 (7.45) | -5.30 (6.50)

16. Secondary Outcome: Change in the Proportion of Days in Which Smoked Compared to Pre-quit Use
Description: Participants will self-report number of days smoked in the past 30 days and this will be compared to self-reported number of days smoked 30 days prior to quit.
Time Frame: 6 month follow-up
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tele-health Mobile Contingency Management Intervention | Tele-health for Alcohol and Smoking Cessation
Number analyzed (Participants) | 30 | 15
days | -9.22 (10.98) | -4.70 (11.50)

17. Secondary Outcome: Number of Participants Who Self-report 7 Day Point Prevalence Abstinence From Smoking
Description: Participants will be asked to report on smoking since two weeks past quit date
Time Frame: 6 week follow-up (i.e., end of treatment visit)
Measure: Count of Participants; unit: Participants
Arm/Group | Tele-health Mobile Contingency Management Intervention | Tele-health for Alcohol and Smoking Cessation
Number analyzed (Participants) | 30 | 15
Participants | 12 | 7

18. Secondary Outcome: Number of Participants Who Self-report 7 Day Point Prevalence Abstinence From Smoking
Description: Participants will be asked to report on smoking since two weeks past quit date
Time Frame: 8 week follow-up (i.e., Session 7, end of monitoring visit)
Measure: Count of Participants; unit: Participants
Arm/Group | Tele-health Mobile Contingency Management Intervention | Tele-health for Alcohol and Smoking Cessation
Number analyzed (Participants) | 30 | 15
Participants | 13 | 9

19. Secondary Outcome: Number of Participants Who Self-report Prolonged Abstinence From Alcohol Use
Description: Participants will be asked to report on alcohol use since two weeks past quit
Time Frame: 8 week follow-up (i.e., Session 7, end of monitoring visit)
Measure: Count of Participants; unit: Participants
Arm/Group | Tele-health Mobile Contingency Management Intervention | Tele-health for Alcohol and Smoking Cessation
Number analyzed (Participants) | 30 | 15
Participants | 13 | 1

20. Secondary Outcome: Number of Participants Who Self-report Prolonged Abstinence From Smoking
Description: Participants will be asked to report on alcohol use since two weeks past quit
Time Frame: 6 week follow-up (i.e., end of treatment visit)
Measure: Count of Participants; unit: Participants
Arm/Group | Tele-health Mobile Contingency Management Intervention | Tele-health for Alcohol and Smoking Cessation
Number analyzed (Participants) | 30 | 15
Participants | 11 | 0

21. Secondary Outcome: Number of Participants Who Self-report Prolonged Abstinence From Smoking
Description: Participants will be asked to report on alcohol use since two weeks past quit
Time Frame: 8 week follow-up (i.e., Session 7, end of monitoring visit)
Measure: Count of Participants; unit: Participants
Arm/Group | Tele-health Mobile Contingency Management Intervention | Tele-health for Alcohol and Smoking Cessation
Number analyzed (Participants) | 30 | 15
Participants | 7 | 0

22. Secondary Outcome: Number of Participants Who Self-report 30 Day Point Prevalence Abstinence From Smoking
Description: Participants will be asked to report on smoking since two weeks past quit date
Time Frame: 6 week follow-up (i.e., end of treatment visit)
Measure: Count of Participants; unit: Participants
Arm/Group | Tele-health Mobile Contingency Management Intervention | Tele-health for Alcohol and Smoking Cessation
Number analyzed (Participants) | 30 | 15
Participants | 2 | 2

23. Secondary Outcome: Number of Participants Who Self-report 30 Day Point Prevalence Abstinence From Smoking
Description: Participants will be asked to report on smoking since two weeks past quit date
Time Frame: 8 week follow-up (i.e., Session 7, end of monitoring visit)
Measure: Count of Participants; unit: Participants
Arm/Group | Tele-health Mobile Contingency Management Intervention | Tele-health for Alcohol and Smoking Cessation
Number analyzed (Participants) | 30 | 15
Participants | 5 | 2

24. Secondary Outcome: Number of Smoking Quit Attempts
Description: Participants will be asked to report the number of quit attempts made since quit date
Time Frame: 6 week follow-up (i.e., end of treatment visit)
Measure: Mean (Standard Deviation); unit: smoking quit attempts
Arm/Group | Tele-health Mobile Contingency Management Intervention | Tele-health for Alcohol and Smoking Cessation
Number analyzed (Participants) | 30 | 15
smoking quit attempts | 2.25 (6.58) | 0.86 (0.38)

25. Secondary Outcome: Number of Smoking Quit Attempts
Description: Participants will be asked to report the number of quit attempts made since quit date
Time Frame: 8 week follow-up (i.e., Session 7, end of monitoring visit)
Measure: Mean (Standard Deviation); unit: smoking quit attempts
Arm/Group | Tele-health Mobile Contingency Management Intervention | Tele-health for Alcohol and Smoking Cessation
Number analyzed (Participants) | 30 | 15
smoking quit attempts | 0.44 (1.03) | 4.11 (9.84)

26. Secondary Outcome: Number of Smoking Quit Attempts
Description: Participants will be asked to report the number of quit attempts made since quit date
Time Frame: 6-month follow-up
Measure: Mean (Standard Deviation); unit: smoking quit attempts
Arm/Group | Tele-health Mobile Contingency Management Intervention | Tele-health for Alcohol and Smoking Cessation
Number analyzed (Participants) | 30 | 15
smoking quit attempts | 2.29 (7.17) | 1.00 (1.64)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for approximately seven months, from informed consent signature to the 6-month follow-up visit, which occurred six months after the substance quit date (session 4).
Arm/Group | Tele-health Mobile Contingency Management Intervention | Tele-health for Alcohol and Smoking Cessation
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/15
Serious Adverse Events (participants affected / at risk) | 2/30 | 0/15
Other Adverse Events (participants affected / at risk) | 6/30 | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tele-health Mobile Contingency Management Intervention (N=30) | Tele-health for Alcohol and Smoking Cessation (N=15)
Hospitalization secondary to burned esophagus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hospitalization secondary to flu (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tele-health Mobile Contingency Management Intervention (N=30) | Tele-health for Alcohol and Smoking Cessation (N=15)
Nausea/diarrhea (Gastrointestinal disorders) | 2 (3) | 0 (0) — Participants reported nausea or diarrhea as a possible side effect of bupropion
Increased stress (Psychiatric disorders) | 1 (2) | 0 (0)
Threat of domestic violence (Psychiatric disorders) | 1 (1) | 0 (0) — Participant left home to avoid domestic violence.
Dental surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Increase in depressed mood (Psychiatric disorders) | 1 (1) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Participant reported skin irritation at nicotine patch placement site.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-03-18): https://cdn.clinicaltrials.gov/large-docs/15/NCT02995915/Prot_SAP_000.pdf
  • Informed Consent Form (2018-09-11): https://cdn.clinicaltrials.gov/large-docs/15/NCT02995915/ICF_001.pdf